CLINICAL TRIAL: NCT07182864
Title: Phase I/II Study of MH004 Ointment in Healthy Adult Volunteers and Participants With Mild to Moderate Atopic Dermatitis
Brief Title: MH004 Ointment in Healthy Adult Volunteers and Participants With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MH004-CP002CN
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Ointments

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Phase I. MH004 (0.1%) in healthy volunteers SAD and MAD (Experimental): SAD and MAD
  Interventions: Drug: MH004 0.1% Ointment
- Phase I: MH004 (0.3%) in healthy volunteers SAD and MAD (Experimental): SAD and MAD
  Interventions: Drug: MH004 0.3% Ointment
- Phase I: MH004 (1.0%) in healthy volunteers SAD and MAD (Experimental): SAD and MAD
  Interventions: Drug: MH004 1.0% Ointment
- Phase I: MH004 (3.0%) in healthy volunteers SAD and MAD (Experimental): SAD and MAD
  Interventions: Drug: MH004 3.0% Ointment
- Phase II. MH004 (0.1%) in Atopic Dermatitis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Atopic Dermatitis
  Interventions: Drug: MH004 0.1% Ointment
- Phase II. MH004 (0.3%) in Atopic Dermatitis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Atopic Dermatitis
  Interventions: Drug: MH004 0.3% Ointment
- Experimental: Phase II. MH004 (1.0%) in Atopic Dermatitis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Atopic Dermatitis
  Interventions: Drug: MH004 1.0% Ointment
- Experimental: Phase II. MH004 (3.0%) in Atopic Dermatitis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Atopic Dermatitis
  Interventions: Drug: MH004 3.0% Ointment
- Phase I. Vehicle Ointment in healthy volunteers SAD and MAD (Placebo Comparator): SAD and MAD
  Interventions: Drug: Vehicle Ointment
- Phase II. Vehicle Ointment in Atopic Dermatitis (Placebo Comparator): 28-Day Repeated Dosing in Participants with Mild to Moderate Atopic Dermatitis
  Interventions: Drug: Vehicle Ointment

INTERVENTIONS:
Drug: MH004 0.1% Ointment — MH004 0.1% ointment applied topically to the affected area as a thin film.
  Arms: Phase I. MH004 (0.1%) in healthy volunteers SAD and MAD; Phase II. MH004 (0.1%) in Atopic Dermatitis
Drug: MH004 0.3% Ointment — MH004 0.3% ointment applied topically to the affected area as a thin film.
  Arms: Phase I: MH004 (0.3%) in healthy volunteers SAD and MAD; Phase II. MH004 (0.3%) in Atopic Dermatitis
Drug: MH004 1.0% Ointment — MH004 1.0% ointment applied topically to the affected area as a thin film.
  Arms: Experimental: Phase II. MH004 (1.0%) in Atopic Dermatitis; Phase I: MH004 (1.0%) in healthy volunteers SAD and MAD
Drug: MH004 3.0% Ointment — MH004 3.0% ointment applied topically to the affected area as a thin film.
  Arms: Experimental: Phase II. MH004 (3.0%) in Atopic Dermatitis; Phase I: MH004 (3.0%) in healthy volunteers SAD and MAD
Drug: Vehicle Ointment — Matching vehicle ointment applied topically to the affected area as a thin film.
  Arms: Phase I. Vehicle Ointment in healthy volunteers SAD and MAD; Phase II. Vehicle Ointment in Atopic Dermatitis

SUMMARY:
This is a Phase I/II Study of MH004 in Healthy Adult Volunteers, participants with Mild to Moderate Atopic Dermatitis.

DETAILED DESCRIPTION:
The study includes 2 parts: The first part (Phase I) is the first-in-human trial of MH004, consisting of a single ascending dose (SAD) study and a multiple ascending dose (MAD) study in healthy volunteers. The second part is a multi-center, randomized, double-Blind, vehicle-controlled phase II study to evaluate the safety, tolerability and PK of MH004 Ointment for AD participants, using defined concentrations of the topical cream based on the PK and safety data in healthy volunteers in Phase I.

ELIGIBILITY:
Inclusion Criteria:

1. Phase I: Adults, age 18 - 70 years old, inclusive. Phase II: Adolescents aged ≥ 12 to 17 years, inclusive. Adults, age 18 - 70 years old, inclusive, at time of screening.
2. Phase II: clinical diagnosis of mild to moderate atopic dermatitis (AD) for at least 6 months prior to Day 1.
3. Phase II: IGA 2 to 3, affected BSA 3% to 20% (excluding scalp) at the baseline visit.
4. Participants who agree to discontinue all agents used to treat AD from screening through the final follow-up visit.

   -

Exclusion Criteria:

1. Unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to baseline.
2. Concurrent conditions and history of other diseases:

   * Immunocompromised.
   * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before Baseline.
   * Active acute bacterial, fungal, or viral skin infection within 1 week before Baseline.
   * Any other concomitant skin disorder, pigmentation, or extensive scarring that, in the opinion of the investigator, may interfere with the evaluation of AD lesions or compromise participant safety.
   * Presence of AD lesions only on the hands or feet without prior history of involvement of other classical areas of involvement such as the face or the folds.
   * Other types of eczema.
3. Clinically significant cardiac disease; new cerebral infarction within 6 months from dosing; malignancies within 5 years from dosing; low hemoglobin; severe renal disease on dialysis; liver disease.
4. Systemic corticosteroids treated within 4 weeks before dosing; immunizations or sedating antihistamines treated within 4 weeks before dosing; other topical treatments for AD within 1 week before dosing.
5. Previously received Janus kinase (JAK) inhibitors, systemic or topical.
6. Ultraviolet light therapy or prolonged exposure to UV radiation within 2 weeks before dosing.
7. Liver function tests: AST or ALT ≥ 2 × ULN; alkaline phosphatase and/or bilirubin > 1.5 × ULN.
8. Pregnant or lactating participants, or those considering pregnancy.
9. Alcohol or drug abuse. -

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-10-08 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence and severity of Treatment-Emergent Adverse Events (Safety and Tolerability) | 1 year
  Assess incidence and severity of treatment-emergent adverse events as determined by CTCAE v5.0 The incidence, nature, and severity of AEs/SAEs including relationship to study treatment from MAD initial study drug administration time of randomization until Day 14 for MAD participants. The incidence, nature, and severity of AEs/SAEs leading to treatment discontinuation from MAD initial study drug administration time of randomisation until Day 7 for MAD participants. Clinically significant changes in laboratory parameters, vital signs, 12-lead ECG, and other safety assessments from initial study drug administration time of randomisation until Day 7 for SAD participants. Clinically significant changes in laboratory parameters, vital signs, 12-lead ECG, and other safety assessments from MAD initial study drug administration time of randomisation until Day 14 for MAD participants.
Phase II: Mean Percentage Change From Baseline in EASI Score at Week 4 in Participants Treated With MH004 Ointment | Baseline and week 4.
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 areas of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.

SECONDARY OUTCOMES:
Phase I: Characterization of Pharmacokinetics (Cmax) of MH004 Ointment in Healthy Volunteers or Participants With Mild to Moderate Atopic Dermatitis | Up to 6 Months
  Maximum drug concentration (Cmax)
Phase II: Mean Percentage Change From Baseline in EASI Score at Week 2 | Baseline, Week 2
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 areas of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.
Percentage of Participants Who Achieve a ≥ 50% or ≥ 75% Improvement From Baseline in EASI (EASI-50 or EASI-75) at Weeks 4 | Baseline, Week 4
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD).
Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of 0 to 1 Who Have an Improvement of ≥ 2 Points From Baseline at Weeks 4 | Baseline, Week 4
  IGA is an assessment scale used to determine severity of atopic dermatitis (AD) and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). An IGA responder was defined as a participant achieving an IGA score of 0 to 1 and an IGA score improvement at least 2 from baseline.
Mean Change From Baseline in the Scoring in Atopic Dermatitis at Week 4 | Baseline, Week 4
  SCORAD is a clinical tool used to assess the severity (range/severity) and subjective signs/symptoms (such as itching/insomnia) of AD. The degree of the lesion was scored using the nine-point method. The severity was determined by grading the severity of six signs (erythema, edema, exudation/scabbing, epidermal exfoliation, lichenification and skin dryness) on a 0-3 subscale. The assessment of each physical sign was scored at the most representative lesion sites. Subjective symptoms were scored using the Visual Analogue Scale (VAS), with 0= no pruritus (or insomnia), and 10= the most severe pruritus (or insomnia). The total score is the sum of 5+7x severity /2+VAS (Symptoms), and the SCORAD score ranges from 0 to 103 points. The higher the score, the more severe the AD.
Number of Participants With At Least One Adverse Event (AEs) and as Per Severity | Up to Week 24
  AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No